CLINICAL TRIAL: NCT02174432
Title: An Open Label Extension Study of the Safety and Anti-Pruritic Efficacy of Nalbuphine HCl ER Tablets in Prurigo Nodularis Patients
Brief Title: Open Label Extension Study of Nalbuphine HCl ER in Patients With Prurigo Nodularis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR03ext; 2013-005628-41 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Prurigo Nodularis; Nodularis Prurigo; Prurigo
Keywords: Itch; Chronic Itch; Nalbupine
MeSH Terms: conditions — Prurigo; Pruritus | interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nalbuphine HCl ER (Experimental): nalbuphine HCl ER
  Interventions: Drug: nalbuphine HCl ER

INTERVENTIONS:
Drug: nalbuphine HCl ER — nalbuphine HCl ER BID for up to 50 weeks
  Other Names: nalbuphine

SUMMARY:
The primary objective of the study is to evaluate the overall safety of nalbuphine HCL ER tablets during a treatment period of up to 50 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed participation in the TR03 study

Exclusion Criteria:

* Medical condition or other factors that in the opinion of the Investigator may interfere with the conduct of the study.
* Subject is a pregnant or lactating female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (1):
- University of Münster, Münster, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nalbuphine HCl ER
Started | 36
Completed | 16
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Nalbuphine HCl ER
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
  Europe | 31
Height [Mean (Standard Deviation); unit: cm] | 172.33 (8.15)
Weight [Mean (Standard Deviation); unit: kg] | 79.68 (16.64)

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence and Nature of Treatment Emergent Adverse Events (TEAEs)
Description: Incidence of adverse events is calculated based on events observed on or after the date of first dose, where incidence is defined as the number of subjects who reported one or more events of a particular adverse event divided by the number of subjects who received at least one dose of investigational product. Overall incidence is the proportion of subjects who had one or more adverse events of any type and nature pertains to the incidence of individual events coded by MedDRA nomenclature. An additional consideration was to evaluate incidence of adverse events by dose achieved but this was not done as subjects achieved a maximum dose during the study that varied and, per protocol, dosing could be modified per the investigator, during the course of this extension to TR03. In addition, TR03EXT involved a dose titration whereas events could have been reported well before a subject achieved some partciular dose level. Consequently, such a presentation would have been impossible to discern.
Time Frame: 50 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nalbuphine HCl ER
Number analyzed (Participants) | 36
Participants | 34

ADVERSE EVENTS:
Time Frame: Adverse events collected beginning with the first date and time of dosing through up to 50 weeks of dosing.
Arm/Group | Nalbuphine HCl ER
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 2/36
Other Adverse Events (participants affected / at risk) | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nalbuphine HCl ER (N=36)
Bradycardia (Cardiac disorders) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Ulnocarpal abutment syndrome (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT02174432/Prot_001.pdf
  • Statistical Analysis Plan (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT02174432/SAP_000.pdf